CLINICAL TRIAL: NCT00513435
Title: A Phase II Study of AZD0530 for Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Saracatinib in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00192; 06-074; CDR0000559632 (Registry Identifier: PDQ (Physician Data Query)); N01CM62206 (NIH); NCT01645618 (obsolete NCT alias); NCT01664468 (obsolete NCT alias)
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2013-08

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — saracatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive saracatinib PO or by PEG tube QD on days 1-56. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: saracatinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: saracatinib — Given PO
  Other Names: AZD0530
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying the how well saracatinib works in treating patients with metastatic or recurrent head and neck cancer. Saracatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the median progression-free survival for patients with advanced or recurrent squamous cell carcinoma of the head and neck (HNSCC) treated with AZD0530 (saracatinib).

SECONDARY OBJEC TIVES:

I. To determine overall survival for patients with advanced or recurrent HNSCC treated with AZD0530.

II. To determine objective response rate for patients with advanced or recurrent HNSCC treated with AZD0530.

III. For patients with accessible tumors, to perform pre and post-treatment biopsies to assess the pharmacodynamic effects of AZD0530 on c-Src and downstream signaling molecules STAT3 and STAT5.

OUTLINE:

Patients receive saracatinib orally (PO) or by percutaneous endoscopic gastrostomy (PEG) tube once daily (QD) on days 1-56. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 12 weeks and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck

  * Persistent, recurrent, or metastatic disease that is not amenable to curative-intent therapy with surgery or radiation
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) ≥ 20 mm with conventional techniques or ≥ 10 mm with spiral computed tomography (CT) scan
* Karnofsky performance status ≥ 60%
* White blood cell (WBC) ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin > 9 g/dL
* Total bilirubin within upper institutional limits of normal (ULN)
* Aspartate aminotransferase (AST) /alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Creatinine within ULN OR creatinine clearance ≥ 60 mL/min
* Patients must agree to use adequate birth control for the duration of study participation and for at least 8 weeks after discontinuation of study drug
* May have received 1 prior cytotoxic chemotherapy regimen for recurrent or metastatic disease

Exclusion Criteria:

* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biological composition to AZD0530
* Urine protein: creatinine ratio ≥ 1.0 OR 24-hour urine protein ≥ 1,000 mg
* QTc prolongation ≥ 480 msecs
* Intercurrent symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* History of myocardial infarction within the past year
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy
* Pulmonary fibrosis ≥ grade 2, pleural effusion (non-malignant) ≥ grade 2, or pneumonitis/pulmonary infiltrates ≥ grade 2
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Use of specifically prohibited cytochrome P450 3A4 (CYP3A4)-active agents or substances

  * Prohibited drugs should be discontinued 7 days prior to the administration of the first dose of AZD0530 and for 7 days following discontinuation of AZD0530
* Patients receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Fury, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 08/22/2006 Protocol Closed to Accrual 07/14/2009 Primary Completion Date 03/08/2011 Recruitment Location is the medical clinic
Groups:
- Treatment (Enzyme Inhibitor Therapy): Patients receive saracatinib 175 mg PO or by PEG tube QD on days 1-56. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Response was determined as inicated in the protocol.
Time Frame: From the start of treatment for up to 12 weeks
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 9
participants
  Stable Disease | 1
  Progression of Disease | 8

2. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier method will be used to estimate overall survival.
Time Frame: Up to 12 weeks
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 9
Days | 180 [27 to 1605]

ADVERSE EVENTS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=9)
Death not assoc w CTCAE term- Sudden death (General disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Inf norm ANC/gr1/2 neut-Cellulitis(skin) (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=9)
Fatigue (asthenia, lethargy, malaise) (Metabolism and nutrition disorders) | 6 (14)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (7)
Nausea (Gastrointestinal disorders) | 4 (4)
AST, SGOT (Renal and urinary disorders) | 4 (4)
Alkaline phosphatase (Renal and urinary disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Epistaxis (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less